CLINICAL TRIAL: NCT05212935
Title: A Surveillance Study on Timing and Coverage Of Rotavirus and MenB Vaccine Co-administration in Campania Region, Italy
Acronym: STORM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Andrea Lo Vecchio, MD, PhD, Assistant Professor, Federico II University
Other Study IDs: 432/21
Record Dates: First submitted 2021-12-21; First posted 2022-01-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Vaccination; Rotavirus Infections; Meningococcal Infections
Keywords: Vaccination coverage; Rotavirus; Meningococcus
MeSH Terms: conditions — Rotavirus Infections; Meningococcal Infections | interventions — Rotavirus Vaccines

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children below 12 months of age receiving vaccines according to the National Vaccination Plan: All children who received vaccination in their first 12 months of life between January 2018 and June 2022 in the Regional Vaccination Centers involved in the study.
  Children will be classified in sub-groups, according to different vaccination schedules (single or co-administration) and order of vaccine uptake.
  Interventions: Biological: Rotavirus Vaccine

INTERVENTIONS:
Biological: Rotavirus Vaccine — administration of the 3 doses of Rotavirus human bovine pentavalent reassortant vaccine

SUMMARY:
A two-phases study will be carried out with the following aims

1. st phase (2018-2020)

   * To investigate the vaccination coverage for Rotavirus vaccine (RV) in Campania Region together with other pediatric vaccinations scheduled in the first 12 months of life: hexavalent, pneumococcal conjugate (PCV), meningococcal B (MenB)
   * To collect data on appropriate timing of the 3 doses of human bovine pentavalent reassortant vaccine (RV5) administration
   * To evaluate the frequency of a co-administration of RV5 with other vaccines scheduled in the first 12 months of life (hexavalent/PCV+RV5, MenB+RV5 vs RV5 alone) and assess the variability in co-administration rates according to RV5 dose
2. nd phase (2020-2022)

   * To investigate the effect of Coronavirus-Disease-19 (COVID-19) pandemic on vaccination coverage in the first year of life, focusing on RV vaccination
   * To investigate the effect of COVID-19 pandemic on timing of vaccine administration in the first year of life, focusing on those vaccines without catch-up vaccination schedule (i.e. RV)

Hypothesis are the following:

* Vaccination coverage and timing of vaccines scheduled in the first year of life are not fully aligned with what is established by the Italian National Prevention Plan 2017-2019
* Co-administration of RV5 and MenB in comparison with other coadministration e.g. hexavalent/PCV is lower
* Co-administration of RV5 and MenB allows to ensure appropriate timing of RV vaccination schedule
* COVID-19 pandemic may have affected the overall vaccination coverage as well as the timing of selected vaccination scheduled in the first year of life, with a more relevant impact on vaccines for whom a catch-up vaccination schedule is not feasible, such as RV immunization.

DETAILED DESCRIPTION:
The study will be carried out in collaboration with eight Vaccination Centers, which are responsible in Italy for the organization and delivery of vaccination as well as for overseeing implementation of vaccinations and monitoring coverage, in four provinces of Campania Region (representative of different regional areas) with the following aims:

* To investigate the vaccination coverage for Rotavirus vaccine (RV) in Campania Region together with other pediatric vaccinations scheduled in the first 12 months of life: hexavalent, pneumococcal conjugate (PCV), meningococcal B (MenB)
* To collect data on appropriate timing of the 3 doses of human bovine pentavalent reassortant vaccine (RV5), which is the most used RV vaccine in Campania Region.
* To evaluate the frequency of a co-administration of RV5 with other vaccines scheduled in the first 12 months of life (hexavalent/PCV+RV5, MenB+RV5 vs RV5 alone) and assess the variability in co-administration rates according to RV5 dose
* To investigate the effect of Coronavirus-Disease-19 (COVID-19) pandemic on vaccination coverage and on timing of vaccine administration in the first year of life, focusing on RV vaccination

The study consists of two parallel phases:

1. First phase aimed at enrolling children who received a vaccine in first 12 months of life between January 2018 and December 2020. These data would provide informative data about the pre-pandemic situation and the impact of restrictive measures against COVID-19 on vaccination.
2. Second phase, enrolling children aged between 6 weeks to 12 months who will enter the national Immunization schedule according to the Italian Immunization Plan up to June 2022 (cohort 2021), in order to investigate a possible role of COVID-19 pandemic and new strategies applied at local level for a catch-up vaccination in the first year of life.

A specific digital dataset will be created to collect data about the number of eligible children who received vaccinations in the territory of each Vaccination Center during the study period. The rough data will be extrapolated by an investigator for each Vaccination province through a single chart reviewing from the regional vaccination database. The regional electronic immunization register is currently used for the entire immunization process (from vaccination call-out, to calculating the vaccination coverage, up to send aggregated data to the Ministry of Health in order to estimate the national vaccination coverage).

The characteristics of each vaccine administered will be recorded (i.e. brand, number of doses) as well as the lass of time between vaccination and possible delay.

Anonymized data obtained by the Regional Registry will be used to analyze vaccination coverage according to age and cohort, timing of administration and frequency and type of co-administration.

Hypothesis are the following:

* Vaccination coverage and timing of vaccines scheduled in the first year of life are not fully aligned with what is established by the Italian National Prevention Plan 2017-2019
* Co-administration of RV5 and MenB in comparison with other coadministration e.g. hexavalent/PCV is lower
* Co-administration of RV5 and MenB allows to ensure appropriate timing of RV vaccination schedule
* COVID-19 pandemic may have affected the overall vaccination coverage as well as the timing of selected vaccination scheduled in the first year of life, with a more relevant impact on vaccines for whom a catch-up vaccination schedule is not feasible, such as RV immunization.

ELIGIBILITY:
Inclusion Criteria:

* all children receiving vaccination according to the Italian National Vaccine Prevention Plan 2017-2019

Exclusion Criteria:

* primary outcomes data missing.

Ages: 6 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children receiving vaccination in their first year of life at one of the Vaccination Centers involved in the study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Overall proportion of children fully immunized for RV and proportion of immunized children in each subgroup | 32 weeks
Proportion of children receiving the first RV5 dose within 12 weeks of age | 32 weeks
Proportion of children completing RV5 schedule within 32 weeks of age | 32 weeks
Proportion of children receiving the co-administration RV5 + MenB | 32 weeks

SECONDARY OUTCOMES:
Proportion of children partially immunized (1 or 2 doses) or not immunized for RV in each subgroup | 32 weeks
Proportion of children receiving RV5 immunization doses alone | 32 weeks
Proportion of children receiving the co-administration of RV5+hexavalent/PCV | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lo Vecchio, MD, PhD, Principal Investigator — Federico II University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Poelaert D, Pereira P, Gardner R, Standaert B, Benninghoff B. A review of recommendations for rotavirus vaccination in Europe: Arguments for change. Vaccine. 2018 Apr 19;36(17):2243-2253. doi: 10.1016/j.vaccine.2018.02.080. Epub 2018 Mar 22. PMID 29576308
- [Background] Lo Vecchio A, Liguoro I, Dias JA, Berkley JA, Boey C, Cohen MB, Cruchet S, Salazar-Lindo E, Podder S, Sandhu B, Sherman PM, Shimizu T, Guarino A. Rotavirus immunization: Global coverage and local barriers for implementation. Vaccine. 2017 Mar 14;35(12):1637-1644. doi: 10.1016/j.vaccine.2017.01.082. Epub 2017 Feb 16. PMID 28216189
- [Background] Foster S. Rotavirus vaccine and intussusception. J Pediatr Pharmacol Ther. 2007 Jan;12(1):4-7. doi: 10.5863/1551-6776-12.1.4. No abstract available. PMID 23055840
- [Background] O'Ryan M, Stoddard J, Toneatto D, Wassil J, Dull PM. A multi-component meningococcal serogroup B vaccine (4CMenB): the clinical development program. Drugs. 2014 Jan;74(1):15-30. doi: 10.1007/s40265-013-0155-7. PMID 24338083
- [Background] DeSilva MB, Haapala J, Vazquez-Benitez G, Daley MF, Nordin JD, Klein NP, Henninger ML, Williams JTB, Hambidge SJ, Jackson ML, Donahue JG, Qian L, Lindley MC, Gee J, Weintraub ES, Kharbanda EO. Association of the COVID-19 Pandemic With Routine Childhood Vaccination Rates and Proportion Up to Date With Vaccinations Across 8 US Health Systems in the Vaccine Safety Datalink. JAMA Pediatr. 2022 Jan 1;176(1):68-77. doi: 10.1001/jamapediatrics.2021.4251. PMID 34617975